CLINICAL TRIAL: NCT02877485
Title: The Effectiveness of Nasal Corticosteroids Versus Placebo in Nasal Obstruction in Patients With Nasal Septal Deviation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sam P. Most, Chief, Division of Facial Plastic and Reconstructive Surgery, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-36535
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Nasal Obstruction
MeSH Terms: conditions — Nasal Obstruction | interventions — Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Triamcinolone acetonide then Ayr spray (Active Comparator): This study arm will start with 6 weeks of therapy with the intranasal steroid, followed by 6 weeks of therapy with a placebo, with a two week washout period in between treatments.
  Interventions: Drug: Triamcinolone Acetonide; Drug: Ayr saline nasal mist
- Ayr spray then triamcinolone acetonide (Active Comparator): This study arm will start with 6 weeks of placebo, followed by 6 weeks of therapy with the intranasal steroid, with a two week washout period in between treatments.
  Interventions: Drug: Triamcinolone Acetonide; Drug: Ayr saline nasal mist

INTERVENTIONS:
Drug: Triamcinolone Acetonide — 2 sprays sprayed to both nostrils daily for 42 days.
  Other Names: Nasacort
Drug: Ayr saline nasal mist — 110mcg (2 sprays) sprayed to both nostrils daily for 42 days.

SUMMARY:
The purpose of this project is to determine if intranasal corticosteroids have an effect on nasal obstruction in patients with nasal septal deviation.

DETAILED DESCRIPTION:
Participants were identified at their initial visit to the Stanford Facial Plastic and Reconstructive Surgery Clinic, an academic referral center, in consultation for nasal obstruction. If eligible and interested in participating, patients provided written informed consent prior to randomization.

Eligible participants were patients over the age of 18 years of age with the presence of nasal septal deviation as identified by physical examination, as well as a baseline NOSE score of 35 or greater. Exclusion criteria included a history of nasal or septal surgery, use of intranasal steroids in the three months preceding enrollment, use of systemic steroids in the six months preceding enrollment, and pregnancy or active breastfeeding at the time of enrollment. In order to maximize generalizability of the study, no medications other than systemic and intranasal steroids were used as exclusion criteria.

All study participants received 6 weeks of therapy with an intranasal steroid spray, Nasacort (Chattem Inc), which consists of the steroid triamcinolone acetonide, as well as 6 weeks of placebo with Ayr saline spray (B.F. Ascher). These two study drugs were packaged identically by a local pharmacist and labelled Drug A and Drug B. Nasacort was selected as the intranasal steroid following pharmacist consultation, as this intranasal steroid is less scented than others and therefore was less likely to be distinguishable from the placebo to participants. Participants were instructed to use both drugs as follows: 1 spray per nostril twice a day. Researchers, statistical analysts, and study participants were blinded to the identity of the two drugs until the conclusion of the study. A duration of 6 weeks per drug was selected based on the most commonly observed insurance requirements seen in our practice. Following unblinding, it was determined that Drug A was the placebo, the saline spray, and Drug B was the test drug, the nasal steroid.

Following completion of both study drugs, patients were offered surgical intervention. If interested and medically cleared for surgery, patients underwent surgery. All surgeries were performed by the senior author and included open septorhinoplasty to address septal deviation, with repair of nasal valve stenosis and inferior turbinate reduction performed in some patients as deemed necessary by the senior author.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18
* NOSE score greater than 55
* Nasal septal deviation on exam

Exclusion Criteria:

* Intranasal steroid use within the last three months
* Current systemic steroid use
* Prior septal surgery
* Individuals who are pregnant or actively breastfeeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam P Most, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sedaghat AR, Busaba NY, Cunningham MJ, Kieff DA. Clinical assessment is an accurate predictor of which patients will need septoplasty. Laryngoscope. 2013 Jan;123(1):48-52. doi: 10.1002/lary.23683. Epub 2012 Nov 20. PMID 23169536
- [Background] Stewart MG, Witsell DL, Smith TL, Weaver EM, Yueh B, Hannley MT. Development and validation of the Nasal Obstruction Symptom Evaluation (NOSE) scale. Otolaryngol Head Neck Surg. 2004 Feb;130(2):157-63. doi: 10.1016/j.otohns.2003.09.016. PMID 14990910
- [Background] Lipan MJ, Most SP. Development of a severity classification system for subjective nasal obstruction. JAMA Facial Plast Surg. 2013 Sep-Oct;15(5):358-61. doi: 10.1001/jamafacial.2013.344. PMID 23846399
- [Background] Teti VP, Akdagli S, Most SP. Cost-effectiveness of Corticosteroid Nasal Spray vs Surgical Therapy in Patients With Severe to Extreme Anatomical Nasal Obstruction. JAMA Facial Plast Surg. 2016 May 1;18(3):165-70. doi: 10.1001/jamafacial.2015.2039. PMID 26747790

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Triamcinolone Acetonide Then Ayr Spray | Ayr Spray Then Triamcinolone Acetonide
Started | 22 | 20
Completed | 22 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Triamcinolone Acetonide Then Ayr Spray | Ayr Spray Then Triamcinolone Acetonide | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 41
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (10.1) | 33.7 (14.4) | 33.0 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 11 | 15 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Nasal Obstruction as Measured by Nasal Obstruction Symptom Evaluation (NOSE) Scores Following Therapy With Treatment (Triamcinolone Acetonide) and Placebo (Ayr Saline Spray)
Description: Nasal Obstruction Symptom Evaluation (NOSE) scale:
  A quality of life (QOL) instrument developed to assess nasal obstruction symptoms in patients undergoing septoplasty. It consists of a 5-item questionnaire, scored on a 5-point (0-4) Likert scale. The raw score ranges from 0-20, which is scaled to a score of 0-100 by multiplying the raw score by 5, where '0' represents 'no problem' and, and '100' represent 'worst problem.'
Time Frame: Pre-spray NOSE score - 6 weeks Post spray NOSE score- 2 weeks washout - Pre spray Pre-spray NOSE score - 6 weeks Post spray NOSE score
Population: Patients requiring nasal surgery for nasal breathing complaints, nasal cosmesis or both.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Triamcinolone Acetonide Then Ayr Spray | Ayr Spray Then Triamcinolone Acetonide
Number analyzed (Participants) | 22 | 20
score on a scale
  Baseline: Pre - spray 1 NOSE score | 69.1 (20.4) | 68.5 (18)
  Post - spray 1 / pre- spray 2 NOSE score | 65.2 (20.7) | 65.8 (20.2)
  Post - spray 2 NOSE score | 64.1 (20.6) | 61.5 (21.8)
Statistical Analysis 1: Comparison: Triamcinolone Acetonide Then Ayr Spray vs Ayr Spray Then Triamcinolone Acetonide; 1) H0: mean change in NOSE score from baseline after in study group 1 = mean change in NOSE score from baseline in study group 2 Power calculation: To detect a 20% difference in NOSE scores with 80% power and a 2-sided alpha level of 0.05 required 20 participants per study group, for a total of 40 participants; Test type: Other; p = 0.7, t-test, 2 sided — Statistical Tests: Independent t-test to assess differences in mean change in NOSE scores when comparing the two study groups, and p<0.05 deemed statistically significant; Mean Difference (Net) = 1.5, 95% CI 2-sided [-6.0 to 8.9] — Change in Mean NOSE score from baseline to post saline versus change in NOSE score from baseline to post intranasal steroid

2. Secondary Outcome: Nasal Obstruction Symptom Evaluation (NOSE) Score Following Surgery in Subset of Patients Who Elect to Undergo Surgery.
Description: as for outcome 1
Time Frame: Postoperative time interval (months): 1-2 , 3-5 , 6-9, 9-12, >12.
Population: Pooled analysis of 35 participants who underwent surgery. Paired t-tests were used to assess differences in mean change in NOSE scores at five post-operative time points compared to baseline NOSE scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Surgery Patients: Participants who underwent surgery
Arm/Group | Surgery Patients
Number analyzed (Participants) | 35
score on a scale
  Baseline NOSE score | 70 (18.9)
  Postoperative period: 1-2 months | 16.2 (20.5)
  Postoperative period:3-5 months | 17.6 (16.5)
  Postoperative period:6-9 months | 17.2 (19.8)
  Postoperative period: 9-12 months | 22.2 (24.9)
  Postoperative period: >12 months | 20 (18.8)
Statistical Analysis 1: Comparison: Surgery Patients; H0: Mean pre- treatment baseline patient NOSE score = Mean post- treatment baseline patient NOSE score; Test type: Other; p < 0.001, Paired t-test — Paired t-tests to assess differences in mean NOSE score when the treatment groups were combined (saline arm+ steroid arm) at five post-operative time intervals compared to the combined preoperative baseline scores. Significance at p<0.05; Mean Difference (Final Values) = -50, Standard Deviation 27.6

ADVERSE EVENTS:
Time Frame: 6 weeks after start of treatment (after drug spray 1). 14 weeks after start of treatment (after drug spray 2)
Description: No adverse events to report
Groups:
- Ayr Spray: Ayr saline nasal mist: 110mcg (2 sprays) sprayed to both nostrils daily for 42 days.
Arm/Group | Triamcinolone Acetonide | Ayr Spray
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/22 | 0/20

LIMITATIONS AND CAVEATS:
The presence and degree of inferior turbinate hypertrophy, the presence of allergic rhinitis, chronic sinusitis, and other forms of nasal mucosal edema, were not assessed or included in analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT02877485/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-04-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT02877485/Prot_SAP_001.pdf